CLINICAL TRIAL: NCT06619366
Title: The Impact of Coach-guided Risk Communication on the Risk of Major Depression: A Randomized Controlled Trial
Brief Title: The Impact of Coach-guided Risk Communication on the Risk of Major Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, JianLi Wang, Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-7208
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Episode; Risk Reduction; Self Efficacy
Keywords: major depressive episode; risk communication; coach-guided; self-help
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: This is an assessor-blinded RCT with two arms. Participants will be recruited from communities across the country, NOT from medical settings. After screening and baseline assessment, participants will be randomized into: (1) intervention, and (2) control group in a 1:1 ratio. Participants in the intervention group will receive the coach-guided PDRC.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The follow-up assessments will be conducted at the PI's telephone interview laboratory. Over the study period, investigators will be blinded to participants' group status. The survey firm interviewers who conduct baseline assessment and randomization, will not be involved in follow-up interviews. The interviewers who conduct the follow-up interviews will not have access to participants' group status. The coaches will not be involved in follow-up assessments. Given our description of study objectives, participants may know their group status. After the 12-month interview, group status will be linked with interview data by study identification numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized depression risk communication (Experimental): The intervention has two integrated components: PDRC and coach-guidance. The PDRC has five sections. The PDRC will be sent to participants by email/mail within two days after the baseline and follow-up assessments.
  The coach will contact the participant within a week after the PDRC is provided by telephone or video conference, depending on participants' preference. The role of the coach is to assist the participant in understanding and interpreting the PDRC, answering their questions, and helping identify self-help strategies that are feasible for the participant; they do not provide psychotherapy. The coaching session will follow the four processes of motivational interview.
  Interventions: Other: coach-guided personalized depression risk communication
- Placebo control (Active Comparator): Participants in the control group will receive their individualized depression risk information. Receiving individualized depression risk information is considered as "control" because: (1) our previous RCT showed that receiving individualized depression risk information caused no psychological harm and was effective in reducing distress and improving function; (2) Receiving depression risk information was used as control in our pilot study; (3) The pilot study suggested that the coach-guided PDRC may be more effective than receiving depression risk information alone.
  Interventions: Other: depression risk information

INTERVENTIONS:
Other: coach-guided personalized depression risk communication — see information in arm description.
  Arms: Personalized depression risk communication
Other: depression risk information — see information in arm description.
  Arms: Placebo control

SUMMARY:
Depression is a highly prevalent and disabling mental health problem. One way of preventing depression is to stop it before it happens through effective self-management. Working with potential users, a coach-guided, personalized depression risk communication tool (PDRC) was developed for sharing information about individualized depression risk, risk profile (risk factors present), potential risk reduction and evidence-based self-help strategies. It is anticipate that the PDRC will greatly motivate users to actively engage in self-help and help seeking, leading to a reduced risk of depression. The proposed study will recruit 500 male and 500 female adults who are at high risk of having depression across Canada, and randomly allocate them into the intervention and control groups. Participants will be followed for 12 months. The data of the trial will allow us to answer the questions: (1) Can the coach-guided PDRC reduce the risk of depression? (2) Does the intervention motivate people to actively engage in evidence-based self-help and help-seeking behaviors? (3) For whom the intervention works best? and (4) what are the costs and potential savings associated with the intervention? If successful, this project will offer a novel and effective tool for early prevention of major depression in the Canadian general population, help us understand how it works and the cost-effectiveness of implementing such a tool in the community from the economic perspective.

DETAILED DESCRIPTION:
Background and importance:

Depression is a highly prevalent and disabling mental health problem. One cost-effective way of reducing the disease burden associated with depression is selective prevention, i.e., identifying individuals who are at high risk of depression, and intervene before it happens. The investigators developed the first sex-specific multivariable risk predictive algorithms (MVRPs) for major depressive episode (MDE) using data from over 10,000 Canadians. Using the MVRP as the foundation and working with future users, the investigators developed a coach-guided personalized depression risk communication tool (PDRC) for sharing information about individualized depression risk, risk profile (risk factors present), potential risk reduction and self-help strategies. It is anticipate that the coach-guided PDRC will greatly motivate users to actively engage in self-help and help-seeking, leading to a reduced risk of depression in the population.

Goals/Research Aims:

The aims of the proposed randomized controlled trial (RCT) are to evaluate the impacts of the coach-guided PDRC on: (1) the risk of MDE at 12 months, (2) self-help and help-seeking behaviors, (3) the severity of depressive symptoms, and to examine (4) the moderation effect by self-efficacy and (5) the cost effectiveness of the coach-guided PDRC.

Methods/Expertise:

The proposed RCT has two arms: (1) intervention group, receiving the coach-guided PDRC; (2) control group, receiving personalized depression risk information. The study population are male and female adults in the community who are at high risk of having an MDE. Because the tools (MVRP) for estimating the risk of having an MDE are sex-specific, the recruitment and the randomization will be conducted in males and females separately. The investigators plan to recruit and follow 500 male and 500 female adults who are at high risk across Canada random digit dialing method and social media and poster advertisement.

The participants will be assessed at baseline, 3- and 12-month to ascertain short-term and mid-term effects. Data will be analyzed in males and females, separately, controlling for the effects of covariates which include gender and gender role related variables. The investigators will examine how the intervention influences the changes in self-help and help seeking behaviors and in depressive symptoms, whether the intervention effect differ by levels of self-efficacy, and if the economic gain exceeds program-related cost. Following the CONSORT guidelines, the investigators will perform both complete case and intent-to-treat analyses based on randomization. The research team has the needed expertise for conducting the proposed RCT, including psychiatry, epidemiology, biostatistics, health economics, risk communication and large RCTs.

The expected outcomes:

In aim 1, it is expected that participants who receive the coach-guided PDRC will have a significantly lower risk of developing MDE over 12 months than those in the control group. It is expected that the intervention will significantly enhance participants' self-help and help-seeking behaviors (aim 2) and reduce depressive symptoms (aim 3). In aim 4, it is expected to observe that the intervention effect is greater in those with higher level of self-efficacy. Finally, the intervention will achieve preferable cost and saving ratio (aim 5). If successful, this coach-guided PDRC can be a novel and cost-effective program for selective prevention of depression in the Canadian general population.

ELIGIBILITY:
Inclusion Criteria:

* no MDE at baseline, or full remission for 2 months for those who had a past MDE (see below the question).
* Aged 18 and 65 years.
* At high risk of MDE based on the depression risk calculators (predicted risk of 6.5%+ for males and 11.2%+ for females), which represent the top two deciles of male and female populations in Canada.
* Agreement to be contacted for follow-up assessments, and
* no language barriers to English or French

Exclusion Criteria:

individuals who

* cannot provide informed consent,
* do not agree to be followed,
* cannot communicate in English and French, or
* report suicide behaviors (score >0 on item 9 of the Patient Health Questionnaire (PHQ-9)).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of major depressive episode cases | 12 months after randomization.
  The proportion of new onset major depressive episode cases measured by the Composite International Diagnostic Interview (CIDI).

SECONDARY OUTCOMES:
Depressive symptom score | 3 and 12 months
  depressive symptom score measured by Patient Health Questionnaire-9. The score ranges between 0 and 27, with a higher score indicating more severe depression.
change in self-help behaviors | 3 and 12 months
  changes in self-help behavioral score measured by the Self-management Strategy Use Scale (SSUS). The SSUS assesses the frequency of using each of the 14 evidence-based self-help strategies. Frequency of use is rated on a 5-category scale. The score ranges between 14 and 70. A higher score indicates more self-help actions.
The percentage of mental health service use | 12 months
  The percentage of reported use of main stream mental health services

OTHER OUTCOMES:
anxiety symptom score | 3 and 12 months
  anxiety symptom score measured by Generalized Anxiety Disorder-7. The score ranges from 0 to 21. A higher score indicates more severe anxiety.
Cost reduction | 12 months
  Sick leave and productivity measured by Health and Work Performance Questionnaire which collects information about number of sick leave days and presenteeism in the past 30 days. The number of sick leave days will be converted into monetary figure to represent cost.

CONTACTS AND LOCATIONS:
Overall Officials: JianLi Wang, PhD, Principal Investigator — Dalhousie University
Locations (1):
- Faculty of Medicine, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the nature of request.

REFERENCES:
- [Derived] Wang J, Feng C, Hajizadeh M, Lesage A. The impact of a coach-guided personalized depression risk communication program on the risk of major depressive episode: study protocol for a randomized controlled trial. BMC Psychiatry. 2024 Dec 18;24(1):916. doi: 10.1186/s12888-024-06393-9. PMID 39696180